CLINICAL TRIAL: NCT04895033
Title: Brain Responses to Contextual Influences on Drinking Decisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: University of Kansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00147117
Record Dates: First submitted 2021-05-12; First posted 2021-05-20 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: The study uses a within-subjects design with all participants completing the no-responsibility and responsibility conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Responsibility vs No Responsibility (Experimental): Within-subjects experimental manipulation of responsibility vs. no-responsibility condition
  Interventions: Behavioral: Responsibility condition

INTERVENTIONS:
Behavioral: Responsibility condition — During the fMRI scan, participants will complete alcohol purchase task paradigm for hypothetical alcohol rewards under two conditions. In the next-day responsibility condition, we will present a vignette describing a drinking scenario in which participants have a significant activity the next day (e.g., a work, family, or academic obligation the next morning) and participants are asked to imagine they are deciding how much they want to drink in this situation. The control condition will use a vignette describing a typical drinking scenario with no explicit responsibilities the next day

SUMMARY:
This study is using functional magnetic resonance imaging (fMRI) to examine brain activity associated with making decisions about drinking alcohol in everyday situations, some of which may involve important activities happening the next day. The secondary aims are to determine whether severity of alcohol-related problems is related to brain activity and alcohol choices and to examine how different areas of the brain interact in connected networks.

DETAILED DESCRIPTION:
The overall objective of this study is to examine brain activity associated with making decisions about drinking alcohol in everyday situations, some of which may involve important activities happening the next day. The secondary aims are to determine whether severity of alcohol-related problems is related to brain activity and alcohol choices and to examine how different areas of the brain interact in connected networks. The study involves two testing sessions -- a baseline interview conducted virtually or in-person, and a MRI scanning session at University of Kansas Medical Center. Participants (N=80, 50% female, age 21-55) are community adults who report drinking alcohol in excess of NIAAA-recommended weekly drinking limits (i.e., heavy drinkers who consume 14/7+ drinks per week for men/women). Participants will complete hypothetical alcohol purchase tasks during the MRI scan with two conditions being examined. A control condition involves a typical drinking situation with no explicit responsibilities. An experimental condition involves a hypothetical situation with important personally-relevant responsibilities the next day (e.g., a presentation at work, an exam, or caregiving responsibilities).

ELIGIBILITY:
Inclusion Criteria:

1. 21-55 years of age;
2. current heavy alcohol drinking in the past three months, as indicated by reporting consumption of 14 or more drinks per week for men or 7 or more drinks per week for women and at least one heavy drinking episode weekly (5+/4+ drinks in a single occasion for males/females);
3. belong to a category with significant responsibilities, such as being currently employed, a current student, or a caregiver with significant responsibilities;
4. speak English;
5. normal or corrected to normal vision and hearing;
6. able to give informed consent.

Exclusion Criteria:

1. currently engaged in treatment or seeking treatment for alcohol-related problems;
2. major psychiatric illness (psychotic disorder, bipolar disorder, post-traumatic stress disorder);
3. Diagnostic and Statistical Manual Version-5 substance use disorder (except nicotine);
4. attending any in-person session with a positive breath alcohol concentration (BrAC > 0.00%);
5. any contraindications for MRI scanning (e.g., metal in body surgically or accidentally including pacemaker, cochlear implants, aneurysm clips, shrapnel, etc.);
6. history of seizures or anti-seizure medication;
7. history of concussion or other significant brain injury;
8. serious medical illness unsuitable for the MRI scanner based on best clinical judgment

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Alcohol demand | During 1 hour MRI scan
  Participants will report how many standard drinks they would consume at varying prices using a hypothetical Alcohol Purchase Task (APT) procedure. The APT is a validated self-report measure of alcohol consumption (in standard drink units) at escalating prices (18 price intervals, ranging from $0 to $80/drink). Responses on APT are analyzed to generate observed and derived indices of alcohol demand, including: intensity (consumption at free price); breakpoint (maximum price for spent for a single drink); Omax (maximum expenditure on alcohol); and Elasticity (proportionate slope of the alcohol demand curve)
Brain activation | During 1 hour MRI scan
  Blood-oxygen-level-dependent (BOLD) activity measured by functional magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Michael Amlung, PhD, Principal Investigator — University of Kansas
Locations (1):
- Cofrin Logan Center for Addiction Research and Treatment, Lawrence, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
After the study is complete, the researchers are encouraged by NIH funding guidelines to deposit de-identified fMRI data and associated baseline data into a public access archive such as NeuroVault, a secure repository where researchers can publicly store and share unthresholded statistical maps, parcellations, and atlases produced by fMRI studies. The investigators will take all necessary steps to ensure that only de-identified data is made publicly available.
Time Frame: Data will be posted at conclusion of study
Access Criteria: Data will be publicly available to researchers who create an account on neurovault.org